CLINICAL TRIAL: NCT06072898
Title: Engaging Mood Brain Circuits With Psilocybin: a Randomized Neuroimaging Trial in Depression
Brief Title: A Randomized Neuroimaging Trial of Psilocybin in Depression
Acronym: EMBRACE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Sean Michael Nestor, Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 5423
Record Dates: First submitted 2023-09-19; First posted 2023-10-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-06

CONDITIONS: Depressive Disorder; Major Depressive Disorder
Keywords: Psilocybin; Neuroimaging; MRI; Depression; Psychotherapy; Psychedelic
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Psilocybin; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: This study will use a 2-group one-way delayed-start (AB/BB) design, with one group receiving placebo at the first visit and the investigational drug at second, and another group receiving the investigational drug at both visits. An interim analysis will be performed after 20 participants have completed the study to assess preliminary efficacy and safety trends.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Staged Active Treatment Arm (Psilocybin-Psilocybin) (Experimental): This group will receive psilocybin (25mg) at the first and second treatment visit, along with supportive psychotherapy.
  Interventions: Drug: Psilocybin; Behavioral: Supportive psychotherapy
- Placebo to Active Delayed-Start Treatment Arm (MCC-Psilocybin) (Experimental): This group will receive microcrystalline cellulose (25mg) at the first treatment visit and psilocybin (25mg) at the second treatment visit, along with supportive psychotherapy.
  Interventions: Drug: Psilocybin; Other: Microcrystalline cellulose; Behavioral: Supportive psychotherapy

INTERVENTIONS:
Drug: Psilocybin — Psilocybin ([3-[2-(dimethylamino)ethyl]-1H-indol-4-yl] dihydrogen phosphate), 25mg PO.
Other: Microcrystalline cellulose — MCC (excipient), 25mg PO.
  Other Names: MCC
  Arms: Placebo to Active Delayed-Start Treatment Arm (MCC-Psilocybin)
Behavioral: Supportive psychotherapy — Supportive psychotherapy in the form of reassurance, integration, and de-escalatory techniques (if needed). Facilitating rapport and a positive environment.

SUMMARY:
The goal of this neuroimaging clinical trial is to test whether psilocybin produces significant immediate changes in functional brain activity in networks associated with mood regulation and depression compared to placebo in patients with depression. The trial aims to determine if psilocybin:

1. Changes connectivity within brain networks associated with mood and depression
2. Changes blood flow in brain regions associated with mood and depression

Participants will be attend two treatment sessions where they receive an oral medication and supportive psychotherapy. At each session, participants will undergo an MRI scan after drug administration but prior to psychotherapy. Participants will be randomly to assigned to one of two groups that will receive, 1) microcrystalline cellulose (25mg) at the first visit and psilocybin (25mg) at the second visit, or 2) psilocybin (25mg) at both visits, respectively. Differences between groups will be compared to understand what effects on brain activity are specific to psilocybin.

ELIGIBILITY:
Inclusion Criteria:

* Able and voluntarily willing to provide written informed consent at the screening visit.
* Over 18 and under 65 years old
* Able to attend all study visits and complete all required assessment tools without assistance or alteration
* Have a responsible individual/caregiver who is able to monitor the participant at home for 24 hours after each treatment visit
* Must have a psychiatrist and/or general practitioner who is able to provide psychiatric follow-up care
* Mini International Neuropsychiatric Interview (MINI)-confirmed diagnosis of depressive disorder, recurrent or single episode, without psychotic features where the duration of the current episode is at least 3 months
* Depression of at least moderate severity as defined by a Hamilton Depression Rating Scale (HAMD-17) score >17

Exclusion Criteria:

* Uncontrolled or insulin-dependent diabetes
* Women who are pregnant (self-report or via urine test), nursing, or planning a pregnancy during the timespan of the study
* History of seizure disorder except for seizures from electroconvulsive therapy and/or febrile seizures in childhood
* History of stroke, recent myocardial infarction (< 1 year from signing of ICF), uncontrolled hypertension (blood pressure > 140/90 mmHg) or clinically significant arrhythmia within 1 year of signing the ICF
* Abnormal and clinically significant results on a physical examination performed within one month of study participation by a general practitioner, vital signs, ECG, or laboratory test at screening
* QTc prolongation on ECG defined by > 450 ms in males and > 460 ms in females in V5 on a 12-lead ECG
* Positive urine drug screen for illicit drugs or drugs of abuse at screening, a week prior to treatment, and during the trial (any positive urine drug test will be reviewed with participants to determine the pattern of use and eligibility will be determined at the investigator's discretion)
* Serial blood counts to achieve a value to meet eligibility -- abnormalities in screening/baseline blood work (complete blood counts, electrolyte panel, etc.) will be reviewed by MD, then repeated serially until abnormalities resolve
* Any symptoms consistent with psychosis
* Any symptoms consistent with hypomania and/or mania as assessed by a psychiatrist
* Other personal circumstances or behavior judged to be incompatible with establishment of rapport or safe exposure to psilocybin
* Current or past history of bipolar I/II disorder, schizophrenia, schizoaffective disorder, psychotic disorder, or delusional disorder as assessed by a structured clinical interview (MINI)
* ≥ 1 suicide attempt in the past year requiring hospitalization, defined using the Columbia Suicide Severity Rating Scale (CSSRS) (Q6 (past year) = "y") and clinical interview with a psychiatrist
* History of substance use and/or alcohol use disorder, of moderate severity or greater, in the past 12 months
* Lifetime history of substance use disorder with a hallucinogen
* Lifetime history of substance-induced psychosis
* Depression secondary to other medical conditions or bipolar I and II disorder
* Family history of a first degree relative with a diagnosis of schizophrenia or a primary psychotic disorder and/or bipolar disorder
* Exposure to psilocybin or any other psychedelic in the past 12 months prior to screening and/or during the current MDE and use of psychedelics, such as ayahuasca/LSD, during the current depressive episode
* A clinical diagnosis of antisocial personality disorder and/or paranoid personality disorder (defined as meeting DSM-5.0 criteria) based on clinical interview and the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at a clinical interview by a psychiatrist
* An active clinical diagnosis of borderline personality disorder as confirmed by the MINI 7.0
* Diagnosis of any mild or major neurocognitive disorder meeting DSM-5 criteria and based on clinical interview/cognitive screening by a psychiatrist
* Current enrolment in an interventional study for depression or participation in such within 30 days of screening
* Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Regional Blood Flow | Up to 3 weeks
  Changes in cerebral blood flow within three a priori-defined brain regions relevant to mood regulation and depression as assessed by arterial spin labeling acutely at expected peak drug concentration during treatment visits.
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Up to 6 weeks
  Changes in the MADRS relative to baseline at study follow-up visits. Higher scores with respect to the MADRS minimum (0) and maximum (60) values represent a worse treatment outcome .

SECONDARY OUTCOMES:
Functional Network Connectivity | Up to 3 weeks
  Changes in voxel-wise functional connectivity within four a priori-defined and established functional networks relevant to mood regulation and depression as assessed by resting state functional magnetic resonance imaging acutely at the time of expected peak drug concentration during treatment visits.
17-item Hamilton Depression Rating Scale (GRID-HAMD-17) | 24 hours
  Baseline grid-version of the 17-item Hamilton Depression Rating Scale score. The GRID-HAMD is a 17-item clinician-administered rating scale designed to assess severity of depressive symptoms. The score range is 0 to 52, with higher score indicating more severe depression .
Incidence of response | up to 6 weeks
  Incidence of response, calculated as the proportion of participants with a response (defined as a ≥ 50% improvement in MADRS total score from Baseline) at at follow-up after psilocybin administration.
Incidence of remission | up to 6 weeks
  Incidence of remission, calculated as the proportion of participants with remission (defined as MADRS total score <11) at week 3 and 6 following the initial psilocybin/niacin administration.
Patient Health Questionnaire 9-item (PHQ-9) | up to 6 weeks
  The PHQ-9 will be collected at baseline as well as week 3 and 6 post-psilocybin administration. The PHQ-9 is a self-rated measure of depressive symptom severity in the past two weeks. Each of the nine items is rated on a Likert scale, ranging from 0 (not at all) to 3 (nearly every day), and summed for a total score between 0 (no symptoms) to 27 (most severe).
16-item Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16) | up to 6 weeks
  The QIDS-SR-16 will be collected at baseline as well as week 3 and 6 post-psilocybin administration. The QIDS-SR-16 is a self-report scale with scores that range from 0 to 27. Higher scores indicate greater depression .
Columbia Suicide Severity Rating Scale (C-SSRS) | up to 6 weeks
  The C-SSRS will be collected at baseline as well as week 3 and 6 post-psilocybin administration. The C-SSRS evaluates suicidal ideation and behaviour. The suicidal ideation score ranges from 0 (no ideation) to 5 (active suicidal ideation with specific plan and intent). Suicidal ideation intensity score ranges from 0 (no ideation) to 25 (most severe). The presence of suicidal behaviour is rated as a binary response; the lethality of previous actual attempts is rated on a scale of 0 (no or very minor physical damage) to 5 (death) and the potential lethality of actual attempts are rated on a scale of 0 (behaviour not likely to result in injury) to 2 (behaviour likely to result in death despite available medical care) .
Brief Psychiatric Rating Scale (BPRS) | up to 6 weeks
  The BPRS will be collected at baseline as well as week 3 and 6 post-psilocybin administration. The BPRS rating scale has 18 items, each item rated on a severity scale of 1 (not present) to 7 (extremely severe). 0 is entered if the item is not assessed.
Sheehan Disability Scale (SDS) | up to 6 weeks
  The SDS will be collected at baseline as well as week 3 and 6 post-psilocybin administration. The SDS total score ranges from 0 to 30, with 0 representing no impairment and 30 representing severe impairment. The last two items of the scale (Days Lost and Days Unproductive) range from 0 to 7 (higher number denotes greater impairment) .
Generalized Anxiety Disorder-7 (GAD-7) | up to 6 weeks
  The GAD-7 will be collected at baseline as well as week 3 and 6 post-psilocybin administration. Scores from 0 ("Not at all") to 3 ("Nearly every day"), and total score ranges from 0 to 21; a higher score denotes greater symptom severity.
Snaith-Hamilton Pleasure Scale (SHAPS) | up to 6 weeks
  The SHAPS will be collected at baseline as well as week 3 and 6 post-psilocybin administration. The SHAPS is rated on a 4-point Likert scale from 0 ("strongly disagree") to 3 ("strongly agree"). Total score ranges from 14 to 56, wherein a higher score indicates greater hedonic capacity (lower anhedonic severity) .
6-Item Clinician Administered Dissociative Symptom Scale (CADSS-6) | up to 6 weeks
  The CADSS-6 is a simplified 6-item scale that will be collected at both treatment visits as well as week 3 and 6 post-psilocybin administration. Responses range from 0 ("not at all") to 4 ("extremely"). Total scores range from 0-24, wherein a higher score indicates greater dissociation.
Montreal Cognitive Assessment (MoCA) | up to 6 weeks
  The MoCA total score will be collected at baseline as well as week 6 (3 weeks after second treatment visit). This is scale is a cognitive screening assessment tool that tests six domains of cognition, with scores ranging from 0-30, wherein a higher score indicates better cognitive performance: 18-25 points ("Mild cognitive impairment"), 10-17 points ("Moderate cognitive impairment"), less than 10 points ("Severe cognitive impairment").
Hopkins Verbal Learning Test-Revised (HVLT-R) | up to 6 weeks
  The revised HVLT-R total Score will be collected at baseline as well as week 6 (3 weeks after second treatment visit). A list learning test that contains 12 nouns that are read to a participant for three consecutive trials. After each trial, a participant is asked to recall the words that were read to them. The number of words recalled on each trial is summed together to produce a total score. The higher total score equates to a better outcome.
CANTAB Rapid Visual Information Processing | up to 6 weeks
  We will use the CANTAB software program for evaluating cognitive domains baseline as well as week 6 (3 weeks after second treatment visit). Sustained attention will be measured by the Rapid Visual Information Processing task. Responses will be scored as the number of responses recorded as having occurred within 1800 milliseconds of the final digit presentation for each of the target sequences, with more responses reflecting better sustained attention.
CANTAB Reaction Time | up to 6 weeks
  We will use the CANTAB software program for evaluating cognitive domains at baseline as well as week 6 (3 weeks after second treatment visit). Psychomotor speed will be measured by the Reaction Time (RTI) task. Simple reaction time will be the outcome of interest, with faster reaction time (lower latency) reflecting better psychomotor speed.
CANTAB Spatial Working Memory | up to 6 weeks
  The CANTAB software program for evaluating cognitive domains is used at baseline as well as week 6 (3 weeks after second treatment visit). Executive function will be measured by the Spatial Working Memory (RTI) task. This is a search task that stresses executive function and spatial working memory, requiring subjects to use heuristic search strategies. A higher score indicates better performance in spatial working memory.
CANTAB One Touch Stockings of Cambridge | up to 6 weeks
  We will use the CANTAB software program for evaluating cognitive domains at baseline as well as week 6 (3 weeks after second treatment visit). Executive function will be measured by the One Touch Stockings of Cambridge (OTS) task. This is a spatial planning task that stresses executive function, requiring subjects to use reordered stacked objects to match a presented pattern. Fewer 'moves' indicates better executive function.
CANTAB Delayed Matching to Sample | up to 6 weeks
  We will use the CANTAB software program for evaluating cognitive domains at baseline as well as week 6 (3 weeks after second treatment visit). Memory will be measured by the Delayed Matching to Sample (DMS) task. This is a memory task that stresses encoding, requiring subjects to remember and differentiate complex patterns when presented after a delay. More correct responses, or greater accuracy, reflects better memory.
CANTAB Paired-Associates Learning | up to 6 weeks
  We will use the CANTAB software program for evaluating cognitive domains at baseline as well as week 6 (3 weeks after second treatment visit). Memory will be measured by the Paired-Associates Learning (PAL) task. This is a memory task =sensitive to changes in functioning of the medial temporal lobe, requiring subjects to remember and identify previous locations of complex patterns when presented after a delay. More correct responses, or greater accuracy, reflects better memory.
CANTAB Emotion Recognition Task | up to 6 weeks
  We will use the CANTAB software program for evaluating cognitive domains at baseline as well as week 6 (3 weeks after second treatment visit). Social/emotional cognition will be assessed by the Emotion Recognition Task (ERT). Subjects are briefly shown faces morphed to display various emotions of varying intensities, and then required to identify the emotion. Better accuracy defined as number of correct responses reflects better emotional cognition.
Revised Mystical Experience Questionnaire (MEQ30) | up to 8 weeks
  The MEQ30 is a validated self-report revised 30-item questionnaire recording elements that comprise the mystical experience. 0 ("none (not at all)") to 5 ("extreme (more than any other time in my life and stronger than 4)"), with a total scoring range from 0 to 150. Higher scores indicate a more profound mystical experience.
Persistent Effects Questionnaire (PEQ) | 24 hours
  The PEQ is a non-validated self-report 145-item questionnaire that describe any changes in the participants' lives that may be attributed to the psilocybin treatment. Comprises of 6 categories with items rated on a 6-point scale from 0 ("none") to 5 ("extreme"). Higher scores indicate a greater magnitude of the persistent effects following their psilocybin experience.

OTHER OUTCOMES:
Blood biomarkers | up to 5 weeks
  Correlation of blood for circulating biomarkers will occur at baseline. Plasma-derived proteins (brain-derived neurotrophic factor, S100Beta, C-reactive protein) will be measured in blood samples collected at the baseline visit and second treatment visit using fluorometric immunoassays and evaluated as predictors of subsequent treatment response as defined above based on MADRS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Nestor, PhD MD FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; Bradley J MacIntosh, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be available 12 months after the end of the trial and initial publication to qualified researchers who provide a sound proposal that is approved by the study principal investigators. Data sharing agreements must adhere to data sharing policies at the Sunnybrook Research Institute. Examples of data sharing can include individual data meta-analyses, and neuroimaging analyses relevant to psilocybin effects. Investigators requesting access to these data should contact the PIs.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The trial protocol will be published, or accepted for publication, in a peer-reviewed journal prior to study initiation and related documents (protocol, ICF, etc) will then be made available. Results will be published in a manuscript as soon as possible after study completion, thereafter this record will be updated to include results. After study completion, IPD will be made available to other researchers who provide a sound proposal and whose uses of the data will adhere to institutional data sharing policies.

REFERENCES:
- [Derived] Poulin JM, Bigford GE, Lanctot KL, Giacobbe P, Schaffer A, Sinyor M, Rabin JS, Masellis M, Singnurkar A, Pople CB, Lipsman N, Husain MI, Rosenblat JD, Cao X, MacIntosh BJ, Nestor SM. Engaging Mood Brain Circuits with Psilocybin (EMBRACE): a study protocol for a randomized, placebo-controlled and delayed-start, neuroimaging trial in depression. Trials. 2024 Jul 3;25(1):441. doi: 10.1186/s13063-024-08268-6. PMID 38956594